CLINICAL TRIAL: NCT05189145
Title: A Prospective Randomized Study of the Impact of Hormonal Monitoring and Progesterone Supplementation Adjustment on Outcome of Programmed Thawed Embryo Transfer Cycles
Brief Title: Hormonal Monitoring and Progesterone Adjustment in Frozen Embryo Transfer Cycles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0201269
Record Dates: First submitted 2021-12-27; First posted 2022-01-12 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2021-12

CONDITIONS: Female Infertility
Keywords: Hormonal monitoring; Frozen embryos; Progesterone; estradiol
MeSH Terms: conditions — Infertility, Female | interventions — Estradiol; Luteinizing Hormone; Progesterone; Suppositories; Dydrogesterone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (control) (Active Comparator): All patients given 8 mg estradiol valerate orally on daily basis for 13 days beginning with the first day of either a spontaneously or induced menstrual cycle. Patients examined using transvaginal ultrasonography on day 13 of exogenous estrogen supplementation to measure endometrial thickness and to detect signs of escape ovulation. In all Patients progesterone supplements in form of two vaginal prontogest suppositories 400 mg each. Transfer of frozen embryo will be done on day 5 after progesterone supplementation.
  Interventions: Drug: estradiol valerate; Diagnostic Test: transvaginal ultrasound examination; Drug: Progesterone 400 Mg Vaginal Suppository
- group II (experimental) (Experimental): All patients given 8 mg estradiol valerate orally on daily basis for 13 days beginning with the first day of either a spontaneously or induced menstrual cycle. Patients examined using transvaginal ultrasonography on day 13 of exogenous estrogen supplementation to measure endometrial thickness and to detect signs of escape ovulation. In all Patients progesterone supplements in form of two vaginal prontogest suppositories 400 mg each. Transfer of frozen embryo will be done on day 5 after progesterone supplementation.
  progesterone (P4) and estradiol assessed and Progesterone supplement adjustments based on serum level of P4 on day of embryo transfer dividing Group II (Cases) into 3 groups:
  * Group II A: If P4 levels < 5ng/dl, one progesterone supplement in form of 100 mg intramuscular injection daily added
  * Group II B: If P4 levels 5-10ng/dl, dydrogesterone three times daily added
  * Group II C: If P4 levels >10ng, continue on 400 mg prontogest suppositories twice daily
  Interventions: Drug: estradiol valerate; Other: Hormonal monitoring progesterone, estradiol, luteinizing hormone; Diagnostic Test: transvaginal ultrasound examination; Drug: Progesterone 400 Mg Vaginal Suppository; Other: Hormonal monitoring progesterone and estradiol; Drug: Progesterone

INTERVENTIONS:
Drug: estradiol valerate — 8mg orally on daily basis for 13 days beginning with the first day of either a spontaneously or induced menstrual cycle then assess by ultrasound
  Other Names: Progenova
Other: Hormonal monitoring progesterone, estradiol, luteinizing hormone — Serum Progesterone, estrogen & LH measured on day 13 after priming endometrium with 8mg estradiol valerate on a daily basis beginning as early as the first day of menstrual cycle.
  Other Names: P4, E2, LH
  Arms: group II (experimental)
Diagnostic Test: transvaginal ultrasound examination — Patients examined using transvaginal ultrasonography on day 13 of exogenous estrogen supplementation to measure endometrial thickness and to detect signs of escape ovulation
Drug: Progesterone 400 Mg Vaginal Suppository — Progesterone supplements given in form of daily two vaginal prontogest suppositories400 mg each
  Other Names: prontogest 400 mg vaginal suppository
Other: Hormonal monitoring progesterone and estradiol — Measuring the serum Progesterone & Estradiol in the early morning on the day of embryo transfer an progesterone supplementation adjusted as follows: Group II A: If P4 levels < 5ng/dl, one 100 mg intramuscular injection daily added, Group II B: If P4 levels 5-10ng/dl, dydrogesterone three times daily added. Group II C: If P4 levels >10ng, continued on 400 mg prontogest suppositories twice daily
  Other Names: P4 and E2
  Arms: group II (experimental)
Drug: Progesterone — group II A: 100 mg intramuscular injection daily Group II B: If P4 levels 5-10ng/dl dydrogesterone added
  Other Names: prontogest Intramuscular injection, duphaston tab
  Arms: group II (experimental)

SUMMARY:
Hormonal monitoring impact on overall pregnancy rate in frozen embryo transfer (FET)cycles and hence progesterone supplement adjustments remain debatable in current literature. This prospective randomized study aims to investigate the effect of monitoring and follow-up of serum progesterone, estradiol & luteinizing hormone (LH) levels and progesterone supplement adjustments on pregnancy outcomes for FET in programmed hormonal replacement therapy cycles in comparison with ultrasound only in control group

DETAILED DESCRIPTION:
Progesterone (P4) is a steroidal hormone that is required for successful embryo implantation and maintenance of the pregnancy in natural cycles, fresh in vitro fertilization cycles, and frozen embryo transfer (FET) cycles. Women undergoing FET in programmed cycle are unable to provide adequate endogenous P4 and require progesterone supplementation to initiate and maintain the secretory endometrium and pregnancy. There has been previous research into luteal phase support in frozen cycles, which has demonstrated that supplementation of progesterone does impact outcome in FET. Despite this evidence for the role of progesterone, there is surprisingly little data on the optimal values for serum P4 during the luteal phase and specifically on the day of embryo transfer in frozen cycles. Following years of a prevalent belief that the higher values of P4 are better, it seems that there may be an optimal window for P4 values during the luteal phase in bovine IVF. Though progesterone levels on the day of transfer have not yet been studied extensively in humans, tailoring the time of transferring a frozen embryo based on serial P4 values rather than cycle day number alone results in higher pregnancy rates. By direct action on the endometrium, a rise of LH might interfere with endometrial receptivity during a FET cycle, in which no pituitary suppression is used. The significance of LH level on the day before addition of progesterone is not yet well defined. The aim of this study is to investigate the effect of monitoring and follow-up of serum progesterone, estradiol & luteinizing hormone levels on day of embryo transfer on pregnancy outcomes for FET in programmed HRT cycles in comparison with ultrasound only in control group and to evaluate the effect of progesterone supplements adjustments depending on serum progesterone levels on day of FET in affecting clinical pregnancy rate.

ELIGIBILITY:
Inclusion Criteria:

1. Age of female patient 42 years or less
2. Normal uterine cavity
3. All embryos are day 5 or day 6 frozen blastocysts

Exclusion Criteria:

1. History of recurrent implantation failure
2. Previously known major thrombophilia factors
3. Non-compliance to given protocol
4. Endometrial thickness < 7mm after 13 days of priming with estradiol valerate
5. pre-existing metabolic diseases (Diabetes Mellitus & Hypertension).

Ages: 20 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 600 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
live birth rate | assessed 26-40 weeks after embryo transfer
  the number of live births (defined as at least one live born after 28 weeks of gestation) divided by the total number of patients who performed pregnancy tests

SECONDARY OUTCOMES:
clinical pregnancy rate | assessed 4 weeks after embryo transfer
  the number of clinical pregnancies (defined as the presence of a gestational sac with positive heart beat detected by transvaginal ultrasound scan 2 weeks after positive pregnancy test) divided by the number of embryo transfer procedures

CONTACTS AND LOCATIONS:
Overall Officials: Sherif Hebisha, phD, Principal Investigator — Alexandria University
Locations (1):
- Infertility Center, Alexandria, Egypt

REFERENCES:
- [Background] Kang HJ. Programmed versus natural frozen embryo transfer: which is the best nest? Fertil Steril. 2018 Sep;110(4):636-637. doi: 10.1016/j.fertnstert.2018.06.020. No abstract available. PMID 30196954
- [Background] Zeilmaker GH, Alberda AT, van Gent I, Rijkmans CM, Drogendijk AC. Two pregnancies following transfer of intact frozen-thawed embryos. Fertil Steril. 1984 Aug;42(2):293-6. doi: 10.1016/s0015-0282(16)48029-5. No abstract available. PMID 6745463
- [Background] Zheng Y, Li Z, Xiong M, Luo T, Dong X, Huang B, Zhang H, Ai J. Hormonal replacement treatment improves clinical pregnancy in frozen-thawed embryos transfer cycles: a retrospective cohort study. Am J Transl Res. 2013 Dec 1;6(1):85-90. eCollection 2013. PMID 24349625
- [Background] Kofinas JD, Blakemore J, McCulloh DH, Grifo J. Serum progesterone levels greater than 20 ng/dl on day of embryo transfer are associated with lower live birth and higher pregnancy loss rates. J Assist Reprod Genet. 2015 Sep;32(9):1395-9. doi: 10.1007/s10815-015-0546-7. Epub 2015 Aug 4. PMID 26238390
- [Background] Dong Z, Sun L, Zhang H, Chen Z, Jian Y. The frozen-thawed embryo transfer timing determined by serum progesterone level: a retrospective follow-up study. Eur J Obstet Gynecol Reprod Biol. 2014 Oct;181:210-3. doi: 10.1016/j.ejogrb.2014.07.012. Epub 2014 Jul 30. PMID 25171265
- [Background] Griesinger G, Weig M, Schroer A, Diedrich K, Kolibianakis EM. Mid-cycle serum levels of endogenous LH are not associated with the likelihood of pregnancy in artificial frozen-thawed embryo transfer cycles without pituitary suppression. Hum Reprod. 2007 Oct;22(10):2589-93. doi: 10.1093/humrep/dem207. Epub 2007 Jul 25. PMID 17652451
- [Background] El-Toukhy T, Taylor A, Khalaf Y, Al-Darazi K, Rowell P, Seed P, Braude P. Pituitary suppression in ultrasound-monitored frozen embryo replacement cycles. A randomised study. Hum Reprod. 2004 Apr;19(4):874-9. doi: 10.1093/humrep/deh183. Epub 2004 Mar 11. PMID 15016780